CLINICAL TRIAL: NCT07019584
Title: Feasibility, Acceptability and Benefits of "Wai Ji Match Fun" Card Games on Cognitive Performance and Psychosocial Wellbeing for People With Intellectual Disabilities
Brief Title: "Wai Ji Match Fun" Card Games for People With Intellectual Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, LIU Karen, Professor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HongKongPU_Match Fun Card Game
Record Dates: First submitted 2025-05-26; First posted 2025-06-13 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-06

CONDITIONS: Adults With Intellectual Disability
Keywords: Card game; intellectual disability; cognition; psychosocial wellbeing; feasibility and acceptability
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Intervention Model Description: one-group repeated-measures design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wai Ji March Fun (Experimental): Groups intervention using game activities with Wai Ji Match Fun cards.
  Interventions: Other: Wai Ji Match Fun card games

INTERVENTIONS:
Other: Wai Ji Match Fun card games — Group intervention using game activities with Wai Ji Match Fun cards. A total of eight group sessions, which last for 60 minutes each, will be conducted once a week for a period of 8 weeks.

SUMMARY:
A new set of card game, Wai Ji Match Fun (WJMF), has been developed by Wai Ji Christian Service (WJCS), a non-governmental organization in Hong Kong, specifically designed for individuals with intellectual disabilities (ID). The game aims to enhance cognitive performance and psychosocial well-being while facilitating daily participation.

DETAILED DESCRIPTION:
This study evaluates the feasibility and acceptability of WJMF for individuals with ID, and its immediate and carry-over impacts on psychosocial well-being and cognitive function. Sixty-four adult participants with mild to moderate ID were recruited for the study. Each participant attends a weekly 60-minute WJMF group program over an 8-week period. Groups of four participants are facilitated by occupational therapists or rehabilitation assistants. Outcome measures include the Personal Wellbeing Index - Intellectual Disability (PWI-ID) (Chinese-Cantonese version), the short version of the Prudhoe Cognitive Function Test (PCFT), attendance rates, and staff feedback on feasibility and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* service users attending residential or day training service units
* aged 18 years or older
* diagnosed with mild or moderate intellectual disability
* able to engage in a 60-minute group session

Exclusion Criteria:

- exhibit disruptive behaviours that could hinder group progress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-11 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Feasibility by measuring the attendance rate | From enrollment to the end of treatment at 8 weeks
  Feasibility by measuring the attendance rate.
Staff acceptability | end of the treatment at 8 weeks
  Acceptability survey collecting staff feedback with questions from 0 (completely disagree) to 10 (completely agree)

SECONDARY OUTCOMES:
The Personal Wellbeing Index - Intellectual Disability (PWI-ID) (Chinese - Cantonese version) (Cummins & Lau, 2005) | Enrollment, one week after the end of treatment, seven weeks after the end of treatment
  An 8-item scale measuring 7 domains in quality of life through interviews. The 8 scales include standard of living, health, life achievement, personal relationships, personal safety, community-connectedness, and future security. Participants rate their well-being using a scale tailored to their abilities: a 0-10-point scale or a system utilising 2, 3, or 5 facial expressions to indicate levels of sadness to happiness.
Prudhoe Cognitive Function Test (PCFT) short version (Tyrer et al., 2010) | Enrollment, one week after the end of treatment, seven weeks after the end of treatment
  A structured interview that has been developed to assess cognitive function in subjects with intellectual disability (Kay et al., 2003). The short version of PCFT consists of six sub-domains: orientation, recall-I, language, praxis, recall-II and calculation (Tyrer et al., 2010), totalling 21 questions. The maximum score for the test is 30.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Liu, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
The project is considering applying for external funding. The IPD can be shared after the funding application announcement and after data collection.